CLINICAL TRIAL: NCT06118385
Title: A Randomised, Double-blind, Placebo-controlled, Phase 1 First-in-human Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Food Effect of Single- and Multiple-ascending Doses of BEN8744 in Healthy Subjects.
Brief Title: Study Investigating the Safety, Tolerability, PK and Food Effect of BEN8744.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BenevolentAI Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BB-8744-1001
Record Dates: First submitted 2023-09-22; First posted 2023-11-07 (Actual); Results first posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteer Study

STUDY DESIGN:
Intervention Model Description: The trial will be in 3 parts: Part A will investigate single ascending oral doses of BEN8744; Part B is a 2-way crossover assessment of the effect of food on the PK of BEN8744; and Part C will investigate multiple ascending oral doses of BEN8744
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Part A Dose 1 (Experimental): Part A Dose 1 Single dose of 2 mg BEN8744
  Interventions: Drug: BEN8744
- Part A Dose 2 (Experimental): Part A Dose 2 Single dose of 6 mg BEN8744
  Interventions: Drug: BEN8744
- Part A Dose 3 (Experimental): Part A Dose 3 Single dose of 20 mg BEN8744
  Interventions: Drug: BEN8744
- Part A Dose 4 (Experimental): Part A Dose 4 Single dose of 60 mg BEN8744
  Interventions: Drug: BEN8744
- Part A Dose 5 (Experimental): Part A Dose 5 Single dose of 100 mg BEN8744
  Interventions: Drug: BEN8744
- Part A Dose 6 (Experimental): Part A Dose 6 Single dose of 120 mg BEN8744
  Interventions: Drug: BEN8744
- Part A placebo (Experimental): Part A placebo Single dose of placebo
  Interventions: Drug: Matching Placebo
- Part B Dose 1 fed (Experimental): Part B Dose 1 Fed Single dose of BEN8744 after high-fat meal (Dose 30mg QD)
  Interventions: Drug: BEN8744
- Part B Dose 1 Fasted (Experimental): Part B Dose 1 Fasted Single dose of BEN8744 after 10 hours fasting (Dose 30mg QD)
  Interventions: Drug: BEN8744
- Part B Dose 2 Fed (Experimental): Part B Dose 2 Fed Single dose of BEN8744 after high-fat meal (Dose 50mg QD)
  Interventions: Drug: BEN8744
- Part B Dose 2 Fasted (Experimental): Part B Dose 2 Fasted Single dose of BEN8744 after 10 hours fasting (Dose 50mg QD)
  Interventions: Drug: BEN8744
- Part C Dose 1 (Experimental): Part C Dose 1 14 daily doses of BEN8744 (Dose 30mg BID)
  Interventions: Drug: BEN8744
- Part C Dose 2 (Experimental): Part C Dose 2 14 daily doses of BEN8744 (Dose 50mg BID)
  Interventions: Drug: BEN8744
- Part C placebo (Experimental): Part C placebo 14 daily doses of placebo
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: BEN8744 — Formulated powder in capsule for oral administration. Supplied as filled Size 0 Swedish Orange capsule. Doses: 2mg, 10mg and 40mg.
  Arms: Part A Dose 1; Part A Dose 2; Part A Dose 3; Part A Dose 4; Part A Dose 5; Part A Dose 6; Part B Dose 1 Fasted; Part B Dose 1 fed; Part B Dose 2 Fasted; Part B Dose 2 Fed; Part C Dose 1; Part C Dose 2
Drug: Matching Placebo — Formulated powder in capsule for oral administration. Supplied as filled Size 0 Swedish Orange capsule. Doses: 2mg, 10mg and 40mg.
  Arms: Part A placebo; Part C placebo

SUMMARY:
BEN8744 is an experimental new medicine for treating inflammatory bowel diseases such as Ulcerative Colitis.

The study will test single and repeated oral doses of BEN8744 or placebo. BEN8744 is a first in human study, so will start with a small dose and the dose will be increased as the study progresses. The goal is to find out its side effects and blood levels when taken by mouth and whether food affects the blood levels.

This is a 3-part study (Parts A, B and C) in up to 108 healthy people, aged 18-65.

Part A, will include up to 64 participants, single doses of BEN8744 or placebo. They'll take about 2 weeks to finish the study, stay on the ward for 4 nights and 5 days in a row and make 2 outpatient visits.

Part B, will include up to 12 participants, single doses of BEN8744 with and without food. They'll take up to 3 weeks to finish the study, stay on the ward for 4 nights and 5 days in a row on 2 occasions, and make 2 outpatient visits.

Part C will include up to 32 participants repeat doses of the BEN8744 or placebo for 14 days. They'll take about 4 weeks to complete the study, stay on the ward for 17 nights and 18 days in a row and make 2 outpatient visits.

DETAILED DESCRIPTION:
This first time in human, study will investigate the safety, tolerability, pharmacokinetics (PK) of BEN8744 after single and multiple ascending oral doses in healthy subjects, in both the fed and fasted state. The results of this study will be used to select doses for subsequent studies in patients. This is an exploratory study in healthy volunteers, with no anticipated therapeutic benefit to the participants; involvement of patients, service users or members of the public in the design of the trial is not appropriate.

Primary objectives Part A: To assess the safety and tolerability of single ascending oral doses of BEN8744 in healthy subjects Part B: To characterise the effect of food on the pharmacokinetic profile of at least 1 dose of BEN8744 Part C: To assess the safety and tolerability of multiple ascending oral doses of BEN8744 in healthy subjects

Secondary objectives Part A: To assess the PK profile of BEN8744 after single oral doses in healthy subjects Part B: To assess the safety and tolerability of a single dose of BEN8744 following high-fat food intake relative to fasting conditions in healthy subjects Part C: To assess the PK profile of BEN8744 after repeated oral doses in healthy subjects

Exploratory objective

Part B (and optional in Part C):

To measure BEN8744 in urine and determine renal clearance in healthy subjects. Exploratory characterisation of BEN8744 and its metabolites in plasma, urine, and faeces.

For part A

* Up to 64 subjects, 5 cohorts + 3 optional, 6 active, 2 placebo.
* Subjects will receive a single dose of BEN8744 or placebo, as capsules, after an overnight fast of at least 10 h.
* At each dose level, 6 subjects will receive BEN8744 and 2 will receive matching placebo in an overall ratio of 3:1.
* The starting dose for Group 1 is 2 mg BEN8744 or placebo. It is intended that subsequent cohorts will receive higher doses. The planned doses are:

A1- 2mg A2- 6mg A3- 20mg A4- 60mg A5- 100mg A6 (optional) - 120mg

For Part B

* Up to 12 subjects, 1 cohorts + 1 optional, 2 sessions fasted/fed.
* Each subject in Part B will have 2 study sessions (Sessions 1 and 2), in which they will receive a single dose of BEN8744, by mouth.
* Each subject will receive BEN8744 after an overnight fast of at least 10 h in one session, and after an FDA high-fat breakfast (1,013 kcal, 59.2 g fat [of which 28.1 g saturated fat) in the other session; the order will be randomised 1:1.
* A subject's doses will be separated by a washout of at least 7 days (or 5 half-lives as determined in Part A, whichever is longer).
* Subjects dosed on the same day may be dosed at intervals of at least 10 min.

For Part C:

* Up 32 subjects, 3 cohorts + 1 optional, 6 active, 2 placebo.
* Each subject will receive daily doses of BEN8744 or placebo, by mouth, for 14 days.
* Doses will be taken once or twice daily in the fasted state, unless emerging data indicate they should be taken in the fed state.
* Part C will not start until at least 3 dose levels have been completed in Part A and may also be conducted in parallel with Part B.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female healthy volunteer in good health
2. Aged 18-65 years
3. Body mass index 18.0-30.9 and weight ≥ 50 kg

Exclusion Criteria:

1. Woman who is pregnant or lactating, or pre-menopausal woman who is sexually active and not using a reliable method of contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denisa Wilkes, Principal Investigator — Hammersmith Medicine Research
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A Placebo: Single dose of placebo capsule(s) matched to active dose
- Part A Dose 1: Single 2 mg dose of BEN8744
- Part A Dose 2: Single 6 mg dose of BEN8744
- Part A Dose 3: Single 20 mg dose of BEN8744
- Part A Dose 4: Single 60 mg dose of BEN8744
- Part A Dose 5: Single 100 mg dose of BEN8744
- Part A Dose 6: Single 120 mg dose of BEN8744
- Part B Dose 1: Single 30 mg dose of BEN8744 administered after 10-hour fast and after high-fat breakfast
- Part B Dose 2: Single 50 mg dose of BEN8744 administered after 10-hour fast and after high-fat breakfast
- Part C Placebo: Placebo capsules matched to active dose twice-daily for 14 days
- Part C Dose 1: 30 mg BEN8744 twice-daily for 14 days
- Part C Dose 2: 50 mg BEN8744 twice-daily for 14 days
Period: Overall Study
Arm/Group | Part A Placebo | Part A Dose 1 | Part A Dose 2 | Part A Dose 3 | Part A Dose 4 | Part A Dose 5 | Part A Dose 6 | Part B Dose 1 | Part B Dose 2 | Part C Placebo | Part C Dose 1 | Part C Dose 2
Started | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 6 | 6
Completed | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 4 | 4 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Out-of-range blood tests | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part B (Both Groups): Dose 1: Single 30 mg dose of BEN8744 administered after 10-hour fast and after high-fat breakfast; Dose 2: Single 50 mg dose of BEN8744 administered after 10-hour fast and after high-fat breakfast
- Total: Total of all reporting groups
Arm/Group | Part A Placebo | Part A Dose 1 | Part A Dose 2 | Part A Dose 3 | Part A Dose 4 | Part A Dose 5 | Part A Dose 6 | Part B (Both Groups) | Part C Placebo | Part C Dose 1 | Part C Dose 2 | Total
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 4 | 6 | 6 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (14.83) | 39.0 (8.44) | 27.8 (4.49) | 32.7 (12.77) | 34.3 (4.13) | 43.0 (13.08) | 31.0 (9.08) | 41.9 (14.30) | 38.5 (9.47) | 38.3 (12.75) | 31.5 (5.89) | 35.9 (4.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 0 | 2 | 1 | 1 | 2 | 4 | 0 | 1 | 2 | 22
  Male | 6 | 3 | 6 | 4 | 5 | 5 | 4 | 8 | 4 | 5 | 4 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 4
  Not Hispanic or Latino | 11 | 6 | 5 | 6 | 5 | 6 | 6 | 12 | 3 | 6 | 6 | 72
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 4 | 0 | 1 | 1 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 3 | 2 | 0 | 2 | 2 | 0 | 1 | 0 | 1 | 14
  White | 7 | 4 | 2 | 4 | 4 | 3 | 2 | 6 | 2 | 5 | 3 | 42
  More than one race | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 5
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 4 | 6 | 6 | 76

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Observer's Assessment of Alertness/Sedation Scale (OAAS/S) (Part A)
Description: The investigator/designee scored the participant's level of alertness on a scale of 0 (absence of response to stimulus) to 5 (readily responsive to the subject's name in a normal tone) in each of 4 components (responsiveness, speech, facial expression, eyes). The composite score corresponds to the lowest score for any component. The sum is the sum of the 4 component scores, ranging from 9 to 20. Positive change in composite score or sum is a better outcome; negative change is a worse outcome.
Time Frame: From Baseline (predose on Day 1) through 72 hours postdose
Measure: Mean (Standard Deviation); unit: score on a scale (change)
Groups:
- Part A Dose 4: Single 60 mg dose BEN8744
Arm/Group | Part A Placebo | Part A Dose 1 | Part A Dose 2 | Part A Dose 3 | Part A Dose 4 | Part A Dose 5 | Part A Dose 6
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
score on a scale (change)
  Composite score (0.25 hour) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Composite score (0.5 hour) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Composite score (1 hour) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Composite score (2 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Composite score (3 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Composite score (4 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Composite score (6 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Composite score (8 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Composite score (24 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Composite score (48 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Composite score (72 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (0.25 hour) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (0.5 hour) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (1 hour) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (2 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (3 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (4 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (6 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (8 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (24 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (48 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (72 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

2. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) (Part A)
Description: The participant graded level of alertness by placing a mark on a linear scale from 0 (very alert) to 100 (very drowsy). Negative change is a better outcome; positive change is a worse outcome.
Time Frame: From Baseline (predose on Day 1) through 72 hours postdose
Measure: Mean (Standard Deviation); unit: mm on a 100-mm line (change)
Arm/Group | Part A Placebo | Part A Dose 1 | Part A Dose 2 | Part A Dose 3 | Part A Dose 4 | Part A Dose 5 | Part A Dose 6
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
mm on a 100-mm line (change)
  Score (0.25 hour) | 1.8 (4.59) | -3.0 (7.29) | 0.5 (4.32) | 3.7 (7.37) | -1.2 (1.94) | -5.8 (7.73) | -5.5 (19.42)
  Score (0.5 hour) | 0.3 (5.80) | 0.5 (12.76) | 3.8 (17.29) | 2.7 (13.98) | 1.0 (3.79) | -2.8 (9.52) | -3.3 (35.30)
  Score (1 hour) | 1.9 (4.64) | -8.2 (13.06) | 14.8 (30.64) | 6.3 (12.86) | 1.8 (7.14) | -2.0 (7.38) | -2.0 (37.83)
  Score (2 hours) | 6.7 (12.03) | -9.3 (12.69) | 6.2 (8.33) | 2.0 (12.93) | 1.3 (5.85) | 0.7 (8.52) | 4.0 (38.76)
  Score (3 hours) | 3.5 (9.11) | -10.3 (22.00) | 3.7 (6.59) | 4.3 (17.20) | -1.2 (6.62) | 3.3 (7.66) | -4.7 (30.69)
  Score (4 hours) | 1.2 (11.44) | -11.2 (14.33) | 3.7 (8.52) | 1.2 (14.66) | -2.3 (4.50) | 6.8 (10.46) | 5.0 (28.87)
  Score (6 hours) | 1.8 (7.00) | -14.3 (15.91) | 3.5 (7.23) | 4.3 (27.98) | 7.0 (19.83) | 1.5 (17.03) | -2.2 (34.74)
  Score (8 hours) | 2.1 (9.58) | 3.7 (30.06) | 0.0 (2.37) | 7.3 (24.36) | -2.2 (7.68) | 8.0 (17.20) | -7.8 (28.53)
  Score (24 hours) | -0.4 (10.32) | -5.7 (10.95) | -1.0 (6.54) | -3.3 (9.83) | 0.5 (8.48) | -2.7 (10.86) | -11.5 (31.86)
  Score (48 hours) | -2.5 (9.99) | -10.3 (11.67) | -2.5 (5.47) | -4.0 (10.30) | -2.0 (8.69) | -6.5 (13.43) | -2.8 (32.46)
  Score (72 hours) | -4.1 (10.30) | -15.7 (16.17) | -2.3 (5.54) | -4.5 (9.59) | -3.7 (7.00) | -9.3 (15.21) | -6.5 (33.41)

3. Primary Outcome: Cmax (PK Part B)
Description: Maximum (peak) plasma concentration. Calculated from plasma concentrations at time points below.
Time Frame: Plasma concentrations measured predose on Day 1 and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose in each of the 2 treatment periods (fasted and fed)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part B Dose 1 Fasted: Single 30 mg dose of BEN8744 after 10-hour fast
- Part B Dose 1 Fed: Single 30 mg dose of BEN8744 after a high-fat breakfast
- Part B Dose 2 Fasted: Single 50 mg dose of BEN8744 after 10-hour fast
- Part B Dose 2 Fed: Single 50 mg dose of BEN8744 after a high-fat breakfast
Arm/Group | Part B Dose 1 Fasted | Part B Dose 1 Fed | Part B Dose 2 Fasted | Part B Dose 2 Fed
Number analyzed (Participants) | 5 | 6 | 5 | 5
ng/mL | 76.7 (41.4) | 88.8 (33.2) | 265 (50.0) | 173 (56.3)

4. Primary Outcome: Tmax (PK Part B)
Description: Time to reach maximum (peak) plasma concentration. Calculated from plasma concentrations at time points below.
Time Frame: as for outcome 3
Measure: Median (Full Range); unit: Hours
Groups:
- Part B Dose 1 Fasted: Single 30 mg dose of BEN8744 after a 10-hour fast
- Part B Dose 1 Fed: Single 30 mg dose of BEN8744 after high-fat breakfast
- Part B Dose 2 Fasted: Single 50 mg dose of BEN8744 after a 10-hour fast
- Part B Dose 2 Fed: Single 50 mg dose of BEN8744 after high-fat breakfast
Arm/Group | Part B Dose 1 Fasted | Part B Dose 1 Fed | Part B Dose 2 Fasted | Part B Dose 2 Fed
Number analyzed (Participants) | 5 | 6 | 5 | 5
Hours | 1.08 [1.00 to 3.00] | 2.02 [1.00 to 3.00] | 1.00 [0.500 to 2.03] | 3.00 [2.02 to 4.00]

5. Primary Outcome: AUC24 (PK Part B)
Description: Area under the plasma concentration-time curve from time 0 to 24 hours postdose. Calculated from plasma concentrations at time points below.
Time Frame: Plasma concentrations measured predose on Day 1 and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, and 24 hours postdose in each of the 2 treatment periods (fasted and fed)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hour/mL
Arm/Group | Part B Dose 1 Fasted | Part B Dose 1 Fed | Part B Dose 2 Fasted | Part B Dose 2 Fed
Number analyzed (Participants) | 5 | 6 | 5 | 5
ng.hour/mL | 227 (25.0) | 332 (25.2) | 721 (47.9) | 666 (54.3)

6. Primary Outcome: AUC72 (PK Part B)
Description: Area under the plasma concentration-time curve from time 0 to 72 hours postdose. Calculated from plasma concentrations at time points below.
Time Frame: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hour/mL
Arm/Group | Part B Dose 1 Fasted | Part B Dose 1 Fed | Part B Dose 2 Fasted | Part B Dose 2 Fed
Number analyzed (Participants) | 5 | 6 | 5 | 5
ng.hour/mL | 229 (24.3) | 335 (26.0) | 723 (48.4) | 669 (54.9)

7. Primary Outcome: AUClast (PK Part B)
Description: Area under the plasma concentration-time curve from time zero to time of last measurable concentration. Calculated from plasma concentrations at time points below.
Time Frame: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hour/mL
Arm/Group | Part B Dose 1 Fasted | Part B Dose 1 Fed | Part B Dose 2 Fasted | Part B Dose 2 Fed
Number analyzed (Participants) | 5 | 6 | 5 | 5
ng.hour/mL | 226 (24.8) | 332 (25.7) | 721 (48.5) | 667 (54.9)

8. Primary Outcome: AUCinf (PK Part B)
Description: Area under the plasma concentration-time curve from time 0 to infinity. Calculated from plasma concentrations at time points below.
Time Frame: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hour/mL
Arm/Group | Part B Dose 1 Fasted | Part B Dose 1 Fed | Part B Dose 2 Fasted | Part B Dose 2 Fed
Number analyzed (Participants) | 5 | 6 | 5 | 5
ng.hour/mL | 228 (24.4) | 335 (26.1) | 723 (48.5) | 669 (55.0)

9. Primary Outcome: t1⁄2 (PK Part B)
Description: Terminal half-life. Calculated from plasma concentrations at time points below.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part B Dose 1 Fasted | Part B Dose 1 Fed | Part B Dose 2 Fasted | Part B Dose 2 Fed
Number analyzed (Participants) | 5 | 6 | 5 | 5
Hours | 4.12 (2.26) | 4.83 (3.67) | 4.23 (5.14) | 3.83 (4.69)

10. Primary Outcome: Terminal Rate Constant (PK Part B)
Description: Calculated from plasma concentrations at time points below.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: /hour
Arm/Group | Part B Dose 1 Fasted | Part B Dose 1 Fed | Part B Dose 2 Fasted | Part B Dose 2 Fed
Number analyzed (Participants) | 5 | 6 | 5 | 5
/hour | 0.210 (0.0956) | 0.217 (0.132) | 0.300 (0.144) | 0.340 (0.173)

11. Primary Outcome: CL/F (PK Part B)
Description: Systemic clearance relative to absolute bioavailability. Calculated from plasma concentrations at time points below.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: L/hour
Groups:
- Part B Dose 2 Fasted: Single 30 mg dose of BEN8744 after 10-hour fast
Arm/Group | Part B Dose 1 Fasted | Part B Dose 1 Fed | Part B Dose 2 Fasted | Part B Dose 2 Fed
Number analyzed (Participants) | 5 | 6 | 5 | 5
L/hour | 135 (33.7) | 92.0 (22.7) | 75.1 (34.3) | 82.3 (36.4)

12. Primary Outcome: VZ/F (PK Part B)
Description: Apparent volume of distribution relative to absolute bioavailability. Calculated from plasma concentrations at time points below.
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Part B Dose 1 Fasted | Part B Dose 1 Fed | Part B Dose 2 Fasted | Part B Dose 2 Fed
Number analyzed (Participants) | 5 | 6 | 5 | 5
L | 846 (582) | 550 (268) | 327 (218) | 310 (186)

13. Primary Outcome: %AUCextrap (PK Part B)
Description: Percentage of AUCinf extrapolated from time of last measurable concentration to infinity. Calculated from plasma concentrations collected at time points below.
Time Frame: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC
Arm/Group | Part B Dose 1 Fasted | Part B Dose 1 Fed | Part B Dose 2 Fasted | Part B Dose 2 Fed
Number analyzed (Participants) | 5 | 6 | 5 | 5
Percentage of AUC | 0.991 (70.2) | 0.638 (73.1) | 0.156 (129.4) | 0.198 (78.0)

14. Primary Outcome: Change From Baseline in Observer's Assessment of Alertness/Sedation Scale (OAAS/S) (Part C)
Description: as for outcome 1
Time Frame: From Baseline (predose on Day 1) through 48 hours postdose
Measure: Mean (Standard Deviation); unit: score on a scale (change)
Arm/Group | Part C Placebo | Part C Dose 1 | Part C Dose 2
Number analyzed (Participants) | 4 | 6 | 6
score on a scale (change)
  Composite score (0.25 hour) | 0 (0) | 0 (0) | 0 (0)
  Composite score (0.5 hour) | 0 (0) | 0 (0) | 0 (0)
  Composite score (1 hour) | 0 (0) | 0 (0) | 0 (0)
  Composite score (2 hours) | 0 (0) | 0 (0) | 0 (0)
  Composite score (3 hours) | 0 (0) | 0 (0) | 0 (0)
  Composite score (4 hours) | 0 (0) | 0 (0) | 0 (0)
  Composite score (6 hours) | 0 (0) | 0 (0) | 0 (0)
  Composite score (8 hours) | 0 (0) | 0 (0) | 0 (0)
  Composite score (24 hours) | 0 (0) | 0 (0) | 0 (0)
  Composite score (48 hours) | 0 (0) | 0 (0) | 0 (0)
  Sum (0.25 hour) | 0 (0) | 0 (0) | 0 (0)
  Sum (0.5 hour) | 0 (0) | 0 (0) | 0 (0)
  Sum (1 hour) | 0 (0) | 0 (0) | 0 (0)
  Sum (2 hours) | 0 (0) | 0 (0) | 0 (0)
  Sum (3 hours) | 0 (0) | 0 (0) | 0 (0)
  Sum (4 hours) | 0 (0) | 0 (0) | 0 (0)
  Sum (6 hours) | 0 (0) | 0 (0) | 0 (0)
  Sum (8 hours) | 0 (0) | 0 (0) | 0 (0)
  Sum (24 hours) | 0 (0) | 0 (0) | 0 (0)
  Sum (48 hours) | 0 (0) | 0 (0) | 0 (0)

15. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) (Part C)
Description: as for outcome 2
Time Frame: From Baseline (predose on Day 1) through 48 hours postdose
Measure: Mean (Standard Deviation); unit: mm on a 100-mm line (change)
Arm/Group | Part C Placebo | Part C Dose 1 | Part C Dose 2
Number analyzed (Participants) | 4 | 6 | 6
mm on a 100-mm line (change)
  Score (0.25 hour) | 1.0 (3.56) | 2.2 (13.33) | -0.3 (5.96)
  Score (0.5 hour) | 2.5 (9.29) | 2.7 (14.02) | 1.8 (6.11)
  Score (1 hour) | 27.3 (24.73) | 15.8 (31.91) | 4.0 (15.66)
  Score (2 hours) | 18.8 (24.43) | 13.0 (26.48) | 7.2 (17.85)
  Score (3 hours) | 18.0 (32.14) | 11.0 (30.33) | 7.3 (16.82)
  Score (4 hours) | 15.3 (27.04) | 8.2 (21.03) | 1.5 (9.27)
  Score (6 hours) | 7.3 (22.53) | 5.3 (18.68) | 6.3 (16.43)
  Score (8 hours) | 1.0 (9.63) | 7.3 (18.55) | -2.5 (8.07)
  Score (24 hours) | 25.8 (25.91) | 12.2 (18.36) | 7.2 (24.68)
  Score (48 hours) | 8.0 (6.98) | 3.2 (11.96) | 2.0 (11.37)

16. Primary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS) (Part C)
Description: The C-SSRS is a questionnaire completed by the Investigator, who asks yes/no questions of the participant It I used to categorise risk levels based on the responses.
Time Frame: Completed during screening and on Days 17 and 24
Measure: Count of Participants; unit: Participants
Arm/Group | Part C Placebo | Part C Dose 1 | Part C Dose 2
Number analyzed (Participants) | 4 | 6 | 6
Participants
  No or low risk - Day 17 | 4 | 6 | 6
  No or low risk - Day 24 | 4 | 6 | 6

17. Secondary Outcome: Cmax (PK Part A)
Description: Maximum (peak) plasma concentration. Calculated from plasma concentrations at time points below.
Time Frame: Plasma concentrations measured predose on Day 1 and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: PK analysis conducted with data from participants who received active BEN8774; plasma PK samples from participants in the placebo group were not tested.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A Dose 1 | Part A Dose 2 | Part A Dose 3 | Part A Dose 4 | Part A Dose 5 | Part A Dose 6
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 1.10 (73.9) | 4.20 (77.2) | 43.7 (40.8) | 297 (74.1) | 548 (33.1) | 695 (54.8)

18. Secondary Outcome: Tmax (PK Part A)
Description: Time to reach maximum (peak) plasma concentration. Calculated from plasma concentrations at time points below.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A Dose 1 | Part A Dose 2 | Part A Dose 3 | Part A Dose 4 | Part A Dose 5 | Part A Dose 6
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
Hours | 2.00 [1.98 to 2.05] | 1.50 [0.517 to 3.00] | 2.03 [1.03 to 3.03] | 1.00 [1.00 to 2.00] | 2.00 [1.00 to 3.00] | 1.00 [1.00 to 3.00]

19. Secondary Outcome: AUC24 (PK Part A)
Description: as for outcome 5
Time Frame: Plasma concentrations measured predose on Day 1 and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24 hours postdose
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hour/mL
Arm/Group | Part A Dose 1 | Part A Dose 2 | Part A Dose 3 | Part A Dose 4 | Part A Dose 5 | Part A Dose 6
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng.hour/mL | NA (NA) — The concentration was below the limit of quantitation at some timepoints, resulting in insufficient data to calculate this endpoint. | 13.8 (54.1) | 154 (42.2) | 901 (62.9) | 1781 (40.6) | 1949 (45.1)

20. Secondary Outcome: AUC72 (PK Part A)
Description: as for outcome 6
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hour/mL
Arm/Group | Part A Dose 1 | Part A Dose 2 | Part A Dose 3 | Part A Dose 4 | Part A Dose 5 | Part A Dose 6
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng.hour/mL | NA (NA) — The concentration was below the limit of quantitation at some timepoints, resulting in insufficient data to calculate this endpoint. | 13.9 (54.2) | 155 (42.4) | 904 (63.3) | 1788 (41.1) | 1959 (44.8)

21. Secondary Outcome: AUClast (PK Part A)
Description: Area under the plasma concentration-time curve from time 0 to time of last measurable concentration. Calculated from plasma concentrations at time points below.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hour/mL
Arm/Group | Part A Dose 1 | Part A Dose 2 | Part A Dose 3 | Part A Dose 4 | Part A Dose 5 | Part A Dose 6
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng.hour/mL | 2.56 (76.1) | 12.9 (59.8) | 153 (42.8) | 902 (63.3) | 1786 (41.1) | 1955 (45.0)

22. Secondary Outcome: AUCinf (PK Part A)
Description: as for outcome 8
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hour/mL
Arm/Group | Part A Dose 1 | Part A Dose 2 | Part A Dose 3 | Part A Dose 4 | Part A Dose 5 | Part A Dose 6
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
ng.hour/mL | NA (NA) — The concentration was below the limit of quantitation at some timepoints, resulting in insufficient data to calculate this endpoint. | 13.8 (53.9) | 155 (42.4) | 904 (63.3) | 1788 (41.2) | 1959 (44.8)

23. Secondary Outcome: %AUCextrap (PK Part A)
Description: Percentage of AUCinf extrapolated from time of last measurable concentration to infinity. Calculated from plasma concentrations at time points below.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC
Arm/Group | Part A Dose 1 | Part A Dose 2 | Part A Dose 3 | Part A Dose 4 | Part A Dose 5 | Part A Dose 6
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
Percentage of AUC | 6.62 (NA) — The concentration was below the limit of quantitation at some timepoints, resulting in insufficient data to calculate AUC for all but one participant, so no coefficient of variation can be calculated. | 4.95 (76.2) | 0.910 (69.8) | 0.202 (126.7) | 0.0796 (125.8) | 0.108 (236.0)

24. Secondary Outcome: t1⁄2 (PK Part A)
Description: Terminal half-life. Calculated from plasma concentrations at time points below.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part A Dose 1 | Part A Dose 2 | Part A Dose 3 | Part A Dose 4 | Part A Dose 5 | Part A Dose 6
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
Hours | NA (NA) — The concentration was below the limit of quantitation at some timepoints, resulting in insufficient data to calculate this endpoint. | 1.89 (0.709) | 3.50 (0.983) | 4.51 (3.41) | 5.57 (5.95) | 7.12 (4.48)

25. Secondary Outcome: Terminal Rate Constant (PK Part A)
Description: Calculated from plasma concentrations at time points below.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: /Hour
Arm/Group | Part A Dose 1 | Part A Dose 2 | Part A Dose 3 | Part A Dose 4 | Part A Dose 5 | Part A Dose 6
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
/Hour | NA (NA) — The concentration was below the limit of quantitation at some timepoints, resulting in insufficient data to calculate this endpoint. | 0.419 (0.172) | 0.214 (0.0702) | 0.216 (0.107) | 0.221 (0.127) | 0.143 (0.100)

26. Secondary Outcome: CL/F (PK Part A)
Description: Systemic clearance relative to absolute bioavailability. Calculated from plasma concentrations at time points below.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Part A Dose 1 | Part A Dose 2 | Part A Dose 3 | Part A Dose 4 | Part A Dose 5 | Part A Dose 6
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
L/hour | NA (NA) — The concentration was below the limit of quantitation at some timepoints, resulting in insufficient data to calculate this endpoint. | 489 (287) | 139 (65.5) | 75.0 (36.2) | 59.4 (21.3) | 66.4 (31.2)

27. Secondary Outcome: VZ/F (PK Part A)
Description: as for outcome 12
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Part A Dose 1 | Part A Dose 2 | Part A Dose 3 | Part A Dose 4 | Part A Dose 5 | Part A Dose 6
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
L | NA (NA) — The concentration was below the limit of quantitation at some timepoints, resulting in insufficient data to calculate this endpoint. | 1268 (747) | 666 (241) | 384 (147) | 374 (227) | 720 (549)

28. Secondary Outcome: Change From Baseline in Observer's Assessment of Alertness/Sedation Scale (OAAS/S) (Part B)
Description: as for outcome 1
Time Frame: From Baseline (predose on Day 1) through 72 hours postdose
Measure: Mean (Standard Deviation); unit: score on a scale (change)
Arm/Group | Part B Dose 1 Fasted | Part B Dose 1 Fed | Part B Dose 2 Fasted | Part B Dose 2 Fed
Number analyzed (Participants) | 6 | 6 | 5 | 5
score on a scale (change)
  Composite score (0.25 hour) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Composite score (0.5 hour) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Composite score (1 hour) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Composite score (2 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Composite score (3 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Composite score (4 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Composite score (6 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Composite score (8 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Composite score (24 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Composite score (48 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Composite score (72 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (0.25 hour) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (0.5 hour) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (1 hour) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (2 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (3 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (4 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (6 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (8 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (24 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (48 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Sum (72 hours) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

29. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) (Part B)
Description: as for outcome 2
Time Frame: From Baseline (predose on Day 1) through 72 hours postdose
Measure: Mean (Standard Deviation); unit: mm on a 100-mm line (change)
Arm/Group | Part B Dose 1 Fasted | Part B Dose 1 Fed | Part B Dose 2 Fasted | Part B Dose 2 Fed
Number analyzed (Participants) | 6 | 6 | 5 | 5
mm on a 100-mm line (change)
  Score (0.25 hour) | -0.7 (2.73) | 1.7 (6.80) | -3.0 (4.30) | -1.6 (1.34)
  Score (0.5 hour) | 2.3 (3.78) | 8.0 (12.79) | 3.0 (14.61) | -0.2 (2.86)
  Score (1 hour) | 1.0 (4.10) | 6.2 (12.09) | 16.4 (36.22) | 2.8 (12.56)
  Score (2 hours) | 6.0 (10.94) | 6.7 (14.08) | 14.4 (30.07) | 9.6 (25.44)
  Score (3 hours) | 4.7 (6.92) | 5.0 (17.81) | -2.2 (14.58) | -2.0 (3.39)
  Score (4 hours) | 8.3 (16.54) | 8.3 (10.89) | 2.2 (18.53) | 8.6 (16.06)
  Score (6 hours) | 15.7 (17.51) | 7.0 (19.29) | 10.0 (32.61) | 1.8 (7.98)
  Score (8 hours) | 7.5 (14.87) | 9.8 (15.84) | 1.2 (5.31) | 0.2 (3.42)
  Score (24 hours) | 8.5 (12.18) | 7.7 (11.89) | -6.0 (11.58) | 6.8 (13.14)
  Score (48 hours) | 9.5 (10.84) | 3.5 (9.27) | -5.0 (14.21) | 3.6 (13.28)
  Score (72 hours) | -1.8 (8.33) | 2.3 (9.46) | -6.0 (10.22) | -3.0 (3.32)

30. Secondary Outcome: Cmax (PK Part C)
Description: Maximum (peak) plasma concentration. Calculated from plasma concentrations measured before the morning dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20 and 24 hours after the morning dose on Day 1; before the morning dose on Days 3, 5, 7, 9, 11, and 13; and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20, 24, 36, 48, and 72 hours after the morning dose on Day 14.
Time Frame: Plasma concentrations measured from predose on Day 1 through 72 hours after Day 14 dose (see specific time points above)
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part C Dose 1 | Part C Dose 2
Number analyzed (Participants) | 6 | 6
ng/mL
  AM Day 1 | 77.9 (56.0) | 198 (47.8)
  PM Day 1 | 49.5 (89.2) | 138 (47.8)
  AM Day 14 | 85.4 (50.0) | 241 (49.9)

31. Secondary Outcome: Tmax (PK Part C)
Description: Time to reach maximum (peak) plasma concentration. Calculated from plasma concentrations measured before the morning dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20 and 24 hours after the morning dose on Day 1; before the morning dose on Days 3, 5, 7, 9, 11, and 13; and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20, 24, 36, 48, and 72 hours after the morning dose on Day 14.
Time Frame: as for outcome 30
Population: as for outcome 17
Measure: Median (Full Range); unit: Hours
Arm/Group | Part C Dose 1 | Part C Dose 2
Number analyzed (Participants) | 6 | 6
Hours
  AM Day 1 | 2.00 [0.500 to 2.00] | 1.51 [1.00 to 2.00]
  PM Day 1 | 3.03 [1.00 to 7.95] | 3.00 [2.00 to 4.00]
  AM Day 14 | 2.08 [1.00 to 3.02] | 2.00 [1.00 to 3.00]

32. Secondary Outcome: Ctrough (PK Part C)
Description: Trough plasma concentration. Calculated from plasma concentrations measured before the morning dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20 and 24 hours after the morning dose on Day 1; before the morning dose on Days 3, 5, 7, 9, 11, and 13; and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20, 24, 36, 48, and 72 hours after the morning dose on Day 14.
Time Frame: as for outcome 30
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Part C Dose 1 | Part C Dose 2
Number analyzed (Participants) | 6 | 6
ng/mL
  Day 1, 12 hours | 0.684 [0.385 to 1.22] | 1.65 [0.865 to 3.16]
  Day 2 | 1.81 [0.875 to 3.75] | 3.57 [1.70 to 7.53]
  Day 3 | 2.97 [1.22 to 7.23] | 4.68 [1.78 to 12.3]
  Day 5 | 2.39 [0.978 to 5.83] | 6.47 [2.61 to 16.1]
  Day 7 | 2.73 [1.43 to 5.21] | 7.09 [3.07 to 16.4]
  Day 9 | 2.87 [0.907 to 9.09] | 6.97 [3.63 to 13.4]
  Day 11 | 1.95 [0.647 to 5.90] | 4.27 [2.03 to 9.01]
  Day 13 | 3.41 [1.46 to 7.98] | 4.72 [2.18 to 10.2]
  Day 14 | 3.24 [1.35 to 7.78] | 6.28 [3.34 to 11.8]
  Day 14, 12 hours | 2.19 [1.14 to 4.21] | 4.93 [2.26 to 10.8]

33. Secondary Outcome: AUCtau (PK Part C)
Description: Area under the concentration-time curve across a dosing interval. Calculated from plasma concentrations measured before the morning dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20 and 24 hours after the morning dose on Day 1; before the morning dose on Days 3, 5, 7, 9, 11, and 13; and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20, 24, 36, 48, and 72 hours after the morning dose on Day 14.
Time Frame: as for outcome 30
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hour/mL
Arm/Group | Part C Dose 1 | Part C Dose 2
Number analyzed (Participants) | 6 | 6
ng.hour/mL
  AM Day 1 | 210 (48.3) | 521 (59.2)
  PM Day 1 | 231 (92.5) | 540 (53.9)
  AM Day 14 | 254 (68.9) | 792 (59.0)

34. Secondary Outcome: AUClast (PK Part C)
Description: Area under the concentration-time curve from time 0 to the last measurable timepoint. Calculated from plasma concentrations measured before the morning dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20 and 24 hours after the morning dose on Day 1; before the morning dose on Days 3, 5, 7, 9, 11, and 13; and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20, 24, 36, 48, and 72 hours after the morning dose on Day 14.
Time Frame: as for outcome 30
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hour/mL
Arm/Group | Part C Dose 1 | Part C Dose 2
Number analyzed (Participants) | 6 | 6
ng.hour/mL
  Day1 | 410 (59.0) | 1034 (47.5)
  Day 14 | 270 (67.8) | 831 (59.3)

35. Secondary Outcome: AUC72 (PK Part C)
Description: Area under the plasma concentration-time curve from time 0 to 72 hours postdose. Calculated from plasma concentrations measured at the time points below.
Time Frame: At 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20, 24, 36, 48, and 72 hours after the morning dose on Day 14
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hour/mL
Arm/Group | Part C Dose 1 | Part C Dose 2
Number analyzed (Participants) | 6 | 6
ng.hour/mL | 273 (66.9) | 837 (58.9)

36. Secondary Outcome: t1⁄2 (PK Part C)
Description: Terminal half-life. Maximum (peak) plasma concentration. Calculated from plasma concentrations measured before the morning dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20 and 24 hours after the morning dose on Day 1; before the morning dose on Days 3, 5, 7, 9, 11, and 13; and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20, 24, 36, 48, and 72 hours after the morning dose on Day 14.
Time Frame: as for outcome 30
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part C Dose 1 | Part C Dose 2
Number analyzed (Participants) | 6 | 6
Hours
  Day 1 | 1.68 (0.317) | 1.63 (0.177)
  Day 14 | 5.89 (2.82) | 9.87 (7.35)

37. Secondary Outcome: AUCinf (PK Part C)
Description: Area under the plasma concentration-time curve from time 0 to infinity. Calculated from plasma concentrations measured before the morning dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20 and 24 hours after the morning dose on Day 1; before the morning dose on Days 3, 5, 7, 9, 11, and 13; and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20, 24, 36, 48, and 72 hours after the morning dose on Day 14.
Time Frame: as for outcome 30
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.hour/mL
Arm/Group | Part C Dose 1 | Part C Dose 2
Number analyzed (Participants) | 6 | 6
ng.hour/mL
  Day 1 | 449 (72.3) | 1149 (52.8)
  Day 14 | 273 (66.9) | 839 (58.9)

38. Secondary Outcome: %AUCextrap (PK Part C)
Description: Percentage of AUCinf extrapolated from time of last measurable concentration to infinity. Calculated from plasma concentrations measured before the morning dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20 and 24 hours after the morning dose on Day 1; before the morning dose on Days 3, 5, 7, 9, 11, and 13; and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20, 24, 36, 48, and 72 hours after the morning dose on Day 14.
Time Frame: as for outcome 30
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC
Arm/Group | Part C Dose 1 | Part C Dose 2
Number analyzed (Participants) | 6 | 6
Percentage of AUC
  Day 1 | 1.36 (219.5) | 0.832 (93.4)
  Day 14 | 1.14 (85.3) | 0.921 (63.6)

39. Secondary Outcome: Terminal Rate Constant (PK Part C)
Description: Calculated from plasma concentrations measured before the morning dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20 and 24 hours after the morning dose on Day 1; before the morning dose on Days 3, 5, 7, 9, 11, and 13; and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20, 24, 36, 48, and 72 hours after the morning dose on Day 14.
Time Frame: as for outcome 30
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: /Hour
Arm/Group | Part C Dose 1 | Part C Dose 2
Number analyzed (Participants) | 6 | 6
/Hour
  Day 1 | 0.424 (0.0848) | 0.428 (0.0428)
  Day 14 | 0.169 (0.148) | 0.123 (0.0955)

40. Secondary Outcome: CLSS/F (PK Part C)
Description: Systemic clearance relative to bioavailability at steady state (Day 14). Calculated from plasma concentrations measured at the time points below.
Time Frame: Plasma concentrations measured at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20, 24, 36, 48, and 72 hours after the morning dose on Day 14
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Part C Dose 1 | Part C Dose 2
Number analyzed (Participants) | 6 | 6
L/hour | 139 (87.1) | 70.2 (31.5)

41. Secondary Outcome: VZ/F (PK Part C)
Description: Apparent volume of distribution relative to absolute bioavailability (Day 14). Calculated from plasma concentrations measured before the morning dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20 and 24 hours after the morning dose on Day 1; before the morning dose on Days 3, 5, 7, 9, 11, and 13; and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20, 24, 36, 48, and 72 hours after the morning dose on Day 14.
Time Frame: as for outcome 30
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Part C Dose 1 | Part C Dose 2
Number analyzed (Participants) | 6 | 6
L | 1221 (823) | 977 (874)

42. Secondary Outcome: Rac(AUCtau) (PK Part C)
Description: Area under the concentration-time curve over the dosing interval on Day 14/area under the concentration-time curve over the dosing interval on Day 1 in AM. Calculated from plasma concentrations measured before the morning dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20 and 24 hours after the morning dose on Day 1; before the morning dose on Days 3, 5, 7, 9, 11, and 13; and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20, 24, 36, 48, and 72 hours after the morning dose on Day 14.
Time Frame: as for outcome 30
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part C Dose 1 | Part C Dose 2
Number analyzed (Participants) | 6 | 6
ratio | 1.33 (0.679) | 1.65 (0.840)

43. Secondary Outcome: Rac(Cmax) (PK Part C)
Description: Maximum observed plasma concentration on Day 14/maximum observed plasma concentration on Day 1 in AM. Calculated from plasma concentrations measured before the morning dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20 and 24 hours after the morning dose on Day 1; before the morning dose on Days 3, 5, 7, 9, 11, and 13; and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20, 24, 36, 48, and 72 hours after the morning dose on Day 14.
Time Frame: as for outcome 30
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part C Dose 1 | Part C Dose 2
Number analyzed (Participants) | 6 | 6
ratio | 1.22 (0.673) | 1.29 (0.559)

44. Secondary Outcome: SR(AUC) (PK Part C)
Description: Area under the concentration-time curve across a dosing interval on Day 14/area under the concentration-time curve from time 0 to infinity. Calculated from plasma concentrations measured before the morning dose and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20 and 24 hours after the morning dose on Day 1; before the morning dose on Days 3, 5, 7, 9, 11, and 13; and at 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 12.5, 13, 14, 15, 16, 20, 24, 36, 48, and 72 hours after the morning dose on Day 14.
Time Frame: as for outcome 30
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part C Dose 1 | Part C Dose 2
Number analyzed (Participants) | 6 | 6
ratio | 0.556 (0.275) | 0.733 (0.158)

ADVERSE EVENTS:
Time Frame: From the signing of the informed consent form through 10 days after the last dose (Day 11 in Parts A and B, Day 24 in Part C)
Arm/Group | Part A Placebo | Part A Dose 1 | Part A Dose 2 | Part A Dose 3 | Part A Dose 4 | Part A Dose 5 | Part A Dose 6 | Part B Dose 1 Fasted | Part B Dose 1 Fed | Part B Dose 2 Fasted | Part B Dose 2 Fed | Part C Placebo | Part C Dose 1 | Part C Dose 2
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/5 | 0/4 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/5 | 0/4 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/12 | 1/6 | 1/6 | 4/6 | 2/6 | 2/6 | 1/6 | 1/6 | 1/6 | 0/5 | 2/5 | 3/4 | 1/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Placebo (N=12) | Part A Dose 1 (N=6) | Part A Dose 2 (N=6) | Part A Dose 3 (N=6) | Part A Dose 4 (N=6) | Part A Dose 5 (N=6) | Part A Dose 6 (N=6) | Part B Dose 1 Fasted (N=6) | Part B Dose 1 Fed (N=6) | Part B Dose 2 Fasted (N=5) | Part B Dose 2 Fed (N=5) | Part C Placebo (N=4) | Part C Dose 1 (N=6) | Part C Dose 2 (N=6)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzymes increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/85/NCT06118385/Prot_SAP_000.pdf